CLINICAL TRIAL: NCT01707693
Title: A Lifestyle Physical Activity Intervention for Older Sedentary Women
Acronym: LPAW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 135603
Record Dates: First submitted 2012-10-12; First posted 2012-10-16 (Estimated); Results first posted 2019-10-11 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-09

CONDITIONS: Coronary Heart Disease
Keywords: physical activity; prevention; coronary heart disease; women
MeSH Terms: conditions — Coronary Disease; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle Physical Activity Intervention (Experimental): the women will be randomized to either the LPA Intervention or Information/Attention Comparison groups using a permuted block randomization scheme. Participants in both groups will be followed longitudinally with repeated assessments of LPA (accelerometer & LPA diary), stage of change, and self-efficacy at baseline and 3 and 6 months; and functional health and well-being (SF36) at baseline and 6 months.
  Interventions: Behavioral: Lifestyle Physical Activity Intervention
- Information/Attention Comparison (Active Comparator): the women will be randomized to either the LPA Intervention or Information/Attention Comparison groups using a permuted block randomization scheme. Participants in both groups will be followed longitudinally with repeated assessments of LPA (accelerometer & LPA diary), stage of change, and self-efficacy at baseline and 3 and 6 months; and functional health and well-being (SF36) at baseline and 6 months.
  Interventions: Behavioral: Information / Attention Comparison

INTERVENTIONS:
Behavioral: Lifestyle Physical Activity Intervention — Physical Activity Information given plus Behavioral counseling using motivational interviewing & follow-up
  Arms: Lifestyle Physical Activity Intervention
Behavioral: Information / Attention Comparison — Physical Activity information given & follow-up, no behavioral counseling
  Arms: Information/Attention Comparison

SUMMARY:
Making physical activity an integral part of daily life is imperative to the health and well-being of our nation's older adults. However, no intervention strategy to encourage daily physical activity for older adults, especially older women, has been effective. This feasibility study will test a multi-tailored motivational intervention to increase usual lifestyle physical activity of older sedentary women to reduce their coronary heart disease risks.

DETAILED DESCRIPTION:
Over 98% of older women do not meet national guidelines for physical activity (PA). There is clear evidence that a physically active lifestyle reduces the human and economic cost of heart disease in a dose-response relationship; but current efforts to increase long-term PA in older women are inadequate. The aims of this proposed research are to: 1) determine the feasibility of using an individually tailored motivational counseling intervention method to promote lifestyle physical activity (LPA) in older sedentary women; 2) examine intervention effects by comparing baseline to outcome measures at 3 and 6 months in treatment and information/attention comparison groups; and 3) explore stage of behavior change and self-efficacy and their relationship to LPA, along with functional health.

This will be a single blinded randomized controlled study of sedentary women aged 60 years and older. We will replace "structured aerobic exercise" with lifestyle physical activity (LPA), i.e., self-selected activities performed daily in a purposeful manner to meet the national PA guidelines. A total of 120 older women who are ambulatory and cognitively intact will be recruited from a senior health clinic and randomized to receive either the motivational LPA intervention or information/attention. Women will be assessed at baseline, 3 and 6 months. The theoretically based behavioral intervention is derived from the Transtheoretical Model and other evidence-based physical activity research. We will use a Motivational Interviewing counseling technique delivered by a social worker to individually tailor the LPA intervention to participant preferences, taking into consideration their functional ability and need for information, readiness to change, and self-efficacy. Outcomes of the LPA intervention sessions will include tailored goals and an LPA plan. Intervention participants will also receive the newly developed NIA "Exercise & You" LPA informational booklet with companion digital video disc (DVD) as well as motivational coaching via telephone calls, tapering in frequency for 6 months. The control group will receive the NIA LPA booklet with DVD and attention telephone calls. We will assess changes from baseline in LPA (primary outcome), readiness to change, self-efficacy and function (secondary outcomes) and examine the associations between primary and secondary outcomes in both groups. The allied disciplines of Nursing, Gerontology, Social Work, and Medicine will collaborate to promote PA and cardiovascular health of older women. Undergraduate and graduate student research assistants will contribute to this project. This research has the potential to increase PA of sedentary older women and reduce coronary heart disease risks. If we could increase physical activity in our rapidly growing older population -even modestly, we could make a significant impact to the health of our nation.

ELIGIBILITY:
Inclusion Criteria:

* women > 60 years of age who are Senior Health clinic patients
* health care provider's approval to participate
* ability to speak/read English
* access to a telephone

Exclusion Criteria:

* report participation in a regular physical activity program
* report an unresolved acute illness, such as pneumonia or flu
* fail screening for capacity to provide informed consent
* fail a simple functional screen or are currently nonambulatory
* are unable to complete activities of daily living
* have uncorrectable severe hearing or vision deficits
* have a history of falls in the past 3 months
* have other unforeseen pathology that precludes safe participation

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2012-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leanne L Lefler, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Physical Activity Motivational Interviewing Counseling INTERV: Received educational material on physical activity from the NIH (Physical Activity & You booklet and Go4Life DVD) Received motivational interviewing behavioral counseling intervention times 2 in month Received motivational interviewing counseling and follow-up over the telephone for 6 months, decreasing in frequency.
  This is the active intervention group
- Information/Attention Without Counseling CONTROL: Received informational/educational material on physical activity from the NIH (Physical Activity & You booklet and Go4Life DVD) Received attention phone calls and follow up over 6 months with theme of "overall health" (without counseling).
  This is the Control Group
Period: Overall Study Allocation
Arm/Group | Physical Activity Motivational Interviewing Counseling INTERV | Information/Attention Without Counseling CONTROL
Started (Allocated to Intervention and Control Arms Time 1 measures) | 59 | 62
Completed (Participants that completed both Time 1 (baseline) and Time 2 Measures (3 month)) | 46 | 54
Not Completed | 13 | 8
Not completed — Withdrawal by Subject | 9 | 5
Not completed — Protocol Violation | 4 | 3
Period: Time 3 Measures @ 6 Mth
Arm/Group | Physical Activity Motivational Interviewing Counseling INTERV | Information/Attention Without Counseling CONTROL
Started | 46 | 54
Completed | 46 | 49
Not Completed | 0 | 5
Not completed — Lost to Follow-up | 0 | 3
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Lifestyle Physical Activity Intervention: the women will be randomized to either the LPA Intervention (n=60) or Information/Attention Comparison (I/A, n=60) groups using a permuted block randomization scheme. Participants in both groups will be followed longitudinally with repeated assessments of LPA (accelerometer & LPA diary), stage of change, and self-efficacy at baseline and 3 and 6 months; and functional health and well-being (SF36) at baseline and 6 months.
  Lifestyle Physical Activity Intervention: Behavioral counseling
- Information/Attention Comparison: the women will be randomized to either the LPA Intervention (n=60) or Information/Attention Comparison (I/A, n=60) groups using a permuted block randomization scheme. Participants in both groups will be followed longitudinally with repeated assessments of LPA (accelerometer & LPA diary), stage of change, and self-efficacy at baseline and 3 and 6 months; and functional health and well-being (SF36) at baseline and 6 months.
  Information / Attention Comparison: Information and attention comparison
- Total: Total of all reporting groups
Arm/Group | Lifestyle Physical Activity Intervention | Information/Attention Comparison | Total
Number analyzed (Participants) | 59 | 62 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.9 (6.1) | 68.3 (6.8) | 69.1 (6.5)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 59 | 62 | 121
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 25 | 42
  White | 40 | 37 | 77
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Total Household Yearly Income [Count of Participants; unit: Participants]
  <10K | 4 | 6 | 10
  10-20K | 8 | 10 | 18
  20K-30K | 12 | 11 | 23
  30K-40K | 9 | 9 | 18
  40-50K | 6 | 8 | 14
  >50K | 14 | 16 | 30
  Refused/DK | 6 | 2 | 8
My living status [Count of Participants; unit: Participants]
  Married (live with spouse) | 29 | 29 | 58
  Live alone | 20 | 21 | 41
  Live with children/relative/friend | 10 | 12 | 22
Highest Grade Level [Count of Participants; unit: Participants]
  Grade School | 0 | 0 | 0
  Some HS | 3 | 2 | 5
  HS Graduate/GED | 4 | 10 | 14
  Vocation or Trade School | 1 | 8 | 9
  Some College | 30 | 21 | 51
  College Graduate | 12 | 10 | 22
  Graduate School | 9 | 11 | 20
Number of people in household [Count of Participants; unit: Participants]
  0 | 0 | 3 | 3
  1 | 26 | 27 | 53
  2 | 29 | 28 | 57
  3 | 3 | 3 | 6
  4 | 1 | 0 | 1
  5 | 0 | 1 | 1
Smoker Category [Count of Participants; unit: Participants]
  1_Current Smoker | 3 | 6 | 9
  2_Past Smoker | 20 | 21 | 41
  3_Non-Smoker, with 2nd-Hand Exposure | 25 | 24 | 49
  4_Non-Smoker, without 2nd-Hand Exposure | 11 | 11 | 22
Cardiovascular Disease History [Count of Participants; unit: Participants]
  Yes | 8 | 13 | 21
  No | 51 | 49 | 100
History of High Blood Pressure [Count of Participants; unit: Participants]
  Yes | 44 | 42 | 86
  No | 15 | 20 | 35
History of Diabetes/Borderline Diabetes [Count of Participants; unit: Participants]
  Yes | 15 | 15 | 30
  No | 44 | 47 | 91
Heart Diseases/Angina [Count of Participants; unit: Participants]
  Yes | 6 | 5 | 11
  No | 53 | 57 | 110
Peripheral Vascular Diseases (Poor Circulation) [Count of Participants; unit: Participants]
  Yes | 1 | 7 | 8
  No | 58 | 55 | 113
Kidney or Renal Failure [Count of Participants; unit: Participants]
  Yes | 2 | 0 | 2
  No | 57 | 62 | 119
Stroke [Count of Participants; unit: Participants]
  Yes | 2 | 3 | 5
  No | 57 | 59 | 116
Abdominal Aortic Aneurysm [Count of Participants; unit: Participants]
  Yes | 0 | 1 | 1
  No | 59 | 61 | 120
High Cholesterol [Count of Participants; unit: Participants]
  Yes | 33 | 26 | 59
  No | 26 | 36 | 62
No History of Relevant Issues [Count of Participants; unit: Participants]
  Yes | 9 | 13 | 22
  No | 50 | 49 | 99
Family hx: heart attack or stroke [Count of Participants; unit: Participants]
  Yes | 37 | 37 | 74
  No | 22 | 25 | 47
Family hx: High Blood Pressure [Count of Participants; unit: Participants]
  Yes | 45 | 46 | 91
  No | 14 | 16 | 30
Follows heart-healthy or low fat/sodium diet [Count of Participants; unit: Participants]
  Yes | 23 | 15 | 38
  No | 36 | 47 | 83
Cholesterol check in last 2 years [Count of Participants; unit: Participants]
  Yes | 53 | 60 | 113
  No | 3 | 1 | 4
  DK | 3 | 1 | 4
Currently works outside the home [Count of Participants; unit: Participants]
  Yes | 23 | 15 | 38
  No | 36 | 47 | 83
employment status [Count of Participants; unit: Participants]
  No/Not Answered for 1 | 37 | 47 | 84
  Part time | 12 | 6 | 18
  Full time (40 hours/week) | 10 | 9 | 19
Major provider of care for another person [Count of Participants; unit: Participants]
  Yes | 13 | 10 | 23
  No | 46 | 52 | 98

OUTCOME MEASURES:

1. Primary Outcome: Accelerometer Vector Magnitude Counts
Description: motion data counts calculated from three axes
Time Frame: 3 and 6 months
Population: Number of participants with completed data
Measure: Median (Inter-Quartile Range); unit: Vector Magnitude Counts
Arm/Group | Physical Activity Motivational Interviewing Counseling INTERV | Information/Attention Without Counseling CONTROL
Number analyzed (Participants) | 46 | 54
Vector Magnitude Counts
  3 Months | 345,000 [263,000 to 439,000] | 324,000 [241,000 to 411,000]
  6 months: number analyzed (Participants) | 46 | 49
  6 months | 324,000 [256,000 to 438,000] | 309,000 [243,000 to 364,000]
Statistical Analysis 1: Comparison: Physical Activity Motivational Interviewing Counseling INTERV vs Information/Attention Without Counseling CONTROL; Test type: Superiority — repeated measures mixed model analysis of covariance, with the baseline measurement as a covariate; p = 0.023, ANCOVA — P-value calculated from repeated measures model adjusting for age with a log transformation applied. P-values are one-sided

2. Secondary Outcome: Step of Counts (Per Day)
Description: Number of steps that a person takes per day
Time Frame: 3 and 6 months
Population: Attrition of 5 participants
Measure: Median (Inter-Quartile Range); unit: Steps per day
Arm/Group | Physical Activity Motivational Interviewing Counseling INTERV | Information/Attention Without Counseling CONTROL
Number analyzed (Participants) | 46 | 54
Steps per day
  3 month | 3982 [2787 to 5157] | 3476 [2691 to 4683]
  6 month: number analyzed (Participants) | 46 | 49
  6 month | 3783 [2840 to 4727] | 3160 [2634 to 3891]
Statistical Analysis 1: Comparison: Physical Activity Motivational Interviewing Counseling INTERV vs Information/Attention Without Counseling CONTROL; Test type: Superiority; p = 0.011, ANCOVA — * P-value calculated from repeated measures model adjusting for age with a log transformation applied; * P-value calculated from repeated measures model adjusting for age with a log transformation applied

3. Other Pre Specified Outcome: Self-Efficacy
Description: Self-Efficacy for Exercise Scale used to estimate the strength of self-efficacy beliefs; The tool contains 9 items with an 0-10 answer format from "Not Confident to Very Confident" and summed numerical ratings; higher scores indicate greater self-efficacy.
Time Frame: Baseline, 3mths, 6mths
Population: 8 participants withdrew from the control group and 13 withdrew from the PA intervention at 3 months. At 6 months 5 participants withdrew from the control group and no withdrawals from the PA intervention group
Measure: Mean (Standard Deviation); unit: mean score on a (0-10) scale
Arm/Group | Physical Activity Motivational Interviewing Counseling INTERV | Information/Attention Without Counseling CONTROL
Number analyzed (Participants) | 59 | 62
mean score on a (0-10) scale
  Baseline | 7.8 (2.4) | 7.0 (2.3)
  3-month: number analyzed (Participants) | 46 | 54
  3-month | 7.7 (1.5) | 5.9 (2.1)
  6- month: number analyzed (Participants) | 46 | 49
  6- month | 7.2 (2.3) | 5.9 (2.3)
Statistical Analysis 1: Comparison: Physical Activity Motivational Interviewing Counseling INTERV vs Information/Attention Without Counseling CONTROL; Test type: Other — 2-sided Wilcoxon Rank Sum test; p = 0.033, Wilcoxon (Mann-Whitney)

4. Other Pre Specified Outcome: Stage of Change (SOC)
Description: Exercise Stage of Change information on how ready an individual is to make a change related to participating in physical activity. It consists of four questions (Yes or No response format) in which the individual is rated on current stage of change
Time Frame: Baseline, 3 and 6 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Groups:
- Information/Attention Without Counseling CONTROL: Information/Attention without Counseling CONTROL Received informational/educational material on physical activity from the NIH (Physical Activity & You booklet and Go4Life DVD) Received attention phone calls and follow up over 6 months with theme of "overall health" (without counseling).
  This is the Control Group
Arm/Group | Physical Activity Motivational Interviewing Counseling INTERV | Information/Attention Without Counseling CONTROL
Number analyzed (Participants) | 59 | 62
Participants
  Baseline SOC: Pre-Contemplation | 9 | 7
  Baseline SOC: Contemplation | 1 | 5
  Baseline SOC: Preparation | 48 | 50
  Baseline SOC: Action | 1 | 0
  Baseline SOC: Maintenance | 0 | 0
  3 Month SOC: number analyzed (Participants) | 46 | 54
  3 Month SOC: Pre-Contemplation | 0 | 3
  3 Month SOC: Contemplation | 0 | 1
  3 Month SOC: Preparation | 4 | 17
  3 Month SOC: Action | 36 | 28
  3 Month SOC: Maintenance | 6 | 5
  6 month SOC: number analyzed (Participants) | 46 | 49
  6 month SOC: Pre-Contemplation | 2 | 3
  6 month SOC: Contemplation | 1 | 4
  6 month SOC: Preparation | 2 | 13
  6 month SOC: Action | 0 | 5
  6 month SOC: Maintenance | 41 | 24
Statistical Analysis 1: Comparison: Physical Activity Motivational Interviewing Counseling INTERV vs Information/Attention Without Counseling CONTROL; Test type: Other — counts of stage of change; p = .001, Cochran-Mantel-Haenszel; 2-sided Cochran-Armitage trend test

ADVERSE EVENTS:
Time Frame: From enrollment to 3 months to 6 months
Description: Staff assessed presence of adverse events via regular contact with participants from both study arms throughout the duration of the study.
Groups:
- Physical Activitiy Motiviational Interviewing Counseling INTER: Received educational material on physical activity from the NIH (Physical Activity & You booklet and Go4Life DVD) Received motivational interviewing behavioral counseling intervention times 2 in month Received motivational interviewing counseling and follow-up over the telephone for 6 months, decreasing in frequency.
  This is the active intervention group
Arm/Group | Physical Activitiy Motiviational Interviewing Counseling INTER | Information/Attention Without Counseling CONTROL
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/59 | 1/62
Other Adverse Events (participants affected / at risk) | 0/59 | 0/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Physical Activitiy Motiviational Interviewing Counseling INTER (N=59) | Information/Attention Without Counseling CONTROL (N=62)
Back Injury (Surgical and medical procedures) | 0 (0) | 1 (1) — Patient was diagnosed with L1 compression fracture & underwent vertebroplasty. Past medical history of osteoporosis. Chart review did not support that compression fracture was related to study activities (control group)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes